CLINICAL TRIAL: NCT06757790
Title: Predictors of Primary Ceaseran Section At Women Health Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Mikhail labib melk, Predictors of primary ceaseran section at women health hospital, Assiut University
Other Study IDs: Predictors of ceaseran section
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Highlight the Most Important Preventable Factors That May Help Decrease Rate of Ceaseran Section in Egypt

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary ceaseran section women: A comparison between primary ceaseran section women and primary vaginally delivery women to determine predictors of primary ceaseran section
  Interventions: Other: A comparison between primary ceaseran section women and primary vaginally delivery women to determine predictors of primary ceaseran section
- Primary vaginally delivery women: A comparison between primary ceaseran section women and primary vaginally delivery women to determine predictors of primary ceaseran section
  Interventions: Other: A comparison between primary ceaseran section women and primary vaginally delivery women to determine predictors of primary ceaseran section

INTERVENTIONS:
Other: A comparison between primary ceaseran section women and primary vaginally delivery women to determine predictors of primary ceaseran section — A comparison between primary ceaseran section women and primary vaginally delivery women to determine predictors of primary ceaseran section

SUMMARY:
Predictors of primary Ceaseran section Highlight the most important preventable risk factors that may help decrease rate of ceaseran section in Egypt

DETAILED DESCRIPTION:
A caesarean section is a surgical procedure in which incisions are made through a woman's Anterior abdominal and uterus to deliver the baby. (1) It is performed whenever abnormal conditions are making normal delivery difficult and endangering the life of the mother or the baby. Cesarean section is the most common obstetric surgical procedure worldwide. Although low cesarean delivery rates are associated with an increase in adverse events, higher-than-institution cesarean delivery rates have been shown not to improve maternal or neonatal outcomes but to cause additional costs and unnecessary interventions (2). There is a global concern that the number of cesarean deliveries is increasing worldwide, regardless of health status, age, race, or gestational age. (3) A Cesarean section of can only effectively save the life of mother and child when it is medically justified (4). For mothers or infants who do not require a Cesarean section, there is no advantage to having it. (5) Recently, it has been reported that the rate of cesarean delivery in Egypt is increasing. (6) All women undergoing indicated or voluntary Cesarean section are at risk of various complications and negative consequences for future pregnancies.(7) Therefore, avoiding unnecessary Cesarean section must be a top priority.(8) An increase in Cesarean has been observed to be among women of all ages and race/ethnicities, in every state, and is thought to be due to; decrease in Vaginal Births after Caesarean Section (VBAC), decreased vaginal births of breech presentation, and increased prevalence of high-risk pregnancies such as advanced maternal age and some subjective indications during labour such as non-reassuring fetal status and arrest of dilation

ELIGIBILITY:
a. Inclusion criteria:

1. All pregnant women underwent primary ceaseran section
2. All primiparous women delivered vaginally b. Exclusion criteria:

(1) any women done previous one or more ceaseran section before (2) All pregnant women delivered vaginally before more than one time (2) women had previous uterine scar as hysterectomy, myomectomy (4) any female refused to participate

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study will be conducted at Women's Health Hospital in Assiut University, Department of Obstetrics and Gynecology.
  divided into 2 groups :females had primary ceaseran section for case and primary vaginal delivery for control group
Sampling Method: Non-Probability Sample
Enrollment: 298 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Identify the risk factors of primary ceaseran section | Baseline
  Identify the risk factors of primary ceaseran section and it's predictors among women seeking delivery care in women health hospital

SECONDARY OUTCOMES:
Highlight the most important preventable factors of ceaseran section | Baseline
  Highlight the most important preventable factors that may help decrease rate of ceaseran section in Egypt